CLINICAL TRIAL: NCT06591442
Title: Screening and Prospective Cohort Study of Risk Factors for Enhanced Recovery After Spinal Fusion Surgery in Advanced Age Patient
Status: Enrolling by invitation | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Caoyang, Head of orthopedics; Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: UHCT-IEC-SOP-016-03-01-2024-1; 2024(0735) (Other: Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology)
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lumbar Disk Herniation; Lumbar Spinal Stenosis; Lumbar Spondylolisthesis; Cervical Spondylotic Myelopathy; Cervical Radiculopathy
Keywords: Enhanced recovery after surgery (ERAS); Spinal fusion surgery; Advanced age patient; High risk factors
MeSH Terms: conditions — Intervertebral Disc Displacement; Spinal Stenosis; Spondylolisthesis; Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elderly group patients (60-74 years).
  Interventions: Diagnostic Test: This is an observational study
- Advanced age group patients (≥75 years)
  Interventions: Diagnostic Test: This is an observational study

INTERVENTIONS:
Diagnostic Test: This is an observational study — This study divides the elderly population into two groups: the Elderly group and the Advanced age group. By observing the enhanced recovery after spinal fusion surgery in these two distinct age groups of elderly patients, risk factors affecting postoperative enhanced recovery will be identified. Detection index: Blood routine examination, blood biochemistry, coagulation function, imaging examination (X-ray, CT 3D reconstruction), Japanese Orthopaedic Association (JOA) score, visual analogue scale (VAS) pain score. The number of participants for all adverse events, serious adverse events, implant-related adverse events and drug-related serious adverse events, and the adverse events were summarized accordingly. The severity of adverse events will be rated according to NCI-CTCAE version 4.0.

SUMMARY:
To determine the high risk factors affecting accelerated recovery after spinal fusion surgery in advanced age patient.

DETAILED DESCRIPTION:
To determine the high risk factors affecting accelerated recovery after spinal fusion surgery in elderly patients: a prospective cohort study

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed and dated by subject or guardian
2. Commit to follow the research procedures and cooperate with the whole process of the study
3. The subjects are 60 years old or older, regardless of gender
4. Patients with degenerative spinal diseases requiring spinal fusion surgery
5. Generally in good physical condition
6. Able to adhere to and cooperate with research interventions, such as oral medication
7. In fertile women, contraception should be used for at least one month prior to screening, and they should commit to use contraception throughout the study period and continue until the specified time after the study

Exclusion Criteria:

1. Acute infection
2. Congenital malformation
3. Abnormal anatomy or skeletal variation
4. Malignant tumor
5. The surgical area was locally infected with symptoms of local inflammation
6. Fever or leukocytosis
7. Morbid obesity
8. Pregnant and nursing women
9. Mental illness
10. Acute joint disease, bone resorption, osteopenia and/or osteoporosis. Osteoporosis is a relative contraindication, as this condition may limit the degree of correction that can be produced, the amount of mechanical fixation, and/or the quality of the bone graft
11. Patients who are unwilling to cooperate with post-operative treatment
12. Any time an implant is performed it interferes with the anatomy or intended physiological function of the patient

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Orthopedics, Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, China
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-09-03 (Estimated); Study Completion 2027-09-03 (Estimated)

PRIMARY OUTCOMES:
Safety Metrics for Enhanced Recovery After Spinal Fusion Surgery | Baseline. 7 days, 3 months, 6 months, 9 months and 12 months after surgery
  Blood routine examination, blood biochemistry, coagulation function, imaging examination (X-ray, CT 3D reconstruction). The number of participants for all adverse events, serious adverse events, implant-related adverse events and drug-related serious adverse events, and the adverse events were summarized accordingly. The severity of adverse events will be rated according to NCI-CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedics, Affiliated Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei 430023, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No